CLINICAL TRIAL: NCT04852185
Title: A Cluster-randomised Controlled Phase IV Trial Assessing the Impact of a Vi-Polysaccharide Conjugate Vaccine in Preventing Typhoid Infection in Asante Akim, Ghana (TyVEGHA)
Brief Title: Evaluation of Typhoid Conjugate Vaccine Effectiveness in Ghana
Acronym: TyVEGHA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Kwame Nkrumah University of Science and Technology (Other); University of Cambridge (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Fondation Mérieux (Other); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TyVEGHA2020
Record Dates: First submitted 2021-03-17; First posted 2021-04-21 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Typhoid Fever
Keywords: Typhoid; Typhoid conjugate vaccine; Cluster randomised trial
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Intervention Model Description: Participant- and observer-blinded, cluster-randomised controlled Phase IV trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vi-TT Arm (Experimental): A single dose of Vi-TT to children 9 months to 15 years of age.
  Interventions: Biological: Vi-TT
- MCV-A arm (Active Comparator): A single dose of MCV-A vaccine to the comparator group.
  Interventions: Biological: MCV-A vaccine

INTERVENTIONS:
Biological: Vi-TT — Single-dose V-TT administered to children and adolescents between the ages of 9 months to 15 years.
  Arms: Vi-TT Arm
Biological: MCV-A vaccine — Single-dose of MCV-A vaccine (a meningococcal vaccine)
  Arms: MCV-A arm

SUMMARY:
A cluster-randomised controlled Phase IV trial (cRCT) assessing the impact of a Vi-Polysaccharide conjugate vaccine in preventing typhoid infection in Asante Akim, Ghana (TyVEGHA) with a primary endpoint of determining the total protection conferred by single-dose vaccination with Vi-TT against blood culture-confirmed symptomatic S. Typhi infection in the intervention vaccine clusters, compared with the control vaccine clusters.

DETAILED DESCRIPTION:
Typhoid fever remains a significant health problem in sub-Saharan Africa, with incidence rates >100 cases per 100,000 person-years of observation. Despite the prequalification of safe and effective typhoid conjugate vaccines (TCV), the uptake of these vaccines in African countries has remained low. Real-life effectiveness data, which inform public health programs on the impact of TCVs in reducing typhoid-related mortality and morbidity, are critical to enhancing the introduction of TCVs in high-burden settings. Here we describe a cluster-randomized trial to investigate population-level protection of TCV against blood culture-confirmed typhoid fever. A total of 80 geographically distinct clusters have been delineated within the Agogo district of the Asante Akim region in Ghana. Clusters will be randomized to the intervention arm receiving TCV or a control arm receiving the meningococcal A conjugate vaccine. The primary study endpoint is the overall protection of TCV against blood culture-confirmed typhoid fever. Total, direct, and indirect protection will be measured as secondary outcomes. Blood culture-based enhanced surveillance will enable the estimation of incidence rates in the intervention and control clusters. Evaluation of the real-world impact of TCVs will improve uptake of prequalified/licensed safe and effective typhoid vaccines in public health programs of high burden settings.

ELIGIBILITY:
Inclusion Criteria: In order to be eligible to participate in this study, an individual must meet the following criteria:

* Healthy participants aged 9 months to <16 years (i.e., ≤15 years and 364 days) of age at the time of vaccination
* Participants/Parents/legally authorized representative (LAR) who have voluntarily given informed assent (sought from participants aged 12 years to <16 years) and informed consent
* Participants/Parents/LAR living within study target area at the time of vaccination and willing to follow the study procedures and be available for the entire duration of the study

Exclusion Criteria: An individual who meets any of the following criteria will be excluded from participation in this study:

* Known allergy to any vaccine component
* Self-reported ongoing acute and/or chronic illness
* Any self-reported coagulopathies
* Any medical or social compelling reasons in the judgment of a clinical physician
* Self-reported pregnancy/Positive urine pregnancy test or lactating
* Previous typhoid vaccination in the last 5 years (proven by the presentation of a vaccine card or self-reporting).

Temporary exclusion criteria

* Self-reported fever (elevated tympanic (≥38°C) or axillary temperature (≥37.5°C)) within 24 hours of vaccination
* Self-reported use of antipyretics within 4hours prior to vaccination
* Any other vaccination during the last 4 weeks (proven by the presentation of a vaccine card or self-reporting)
* Girls ≥11 years of age with self-reported irregular menstruation or who do not know their last menstruation date

Ages: 9 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23000 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Protection | 3 years
  The incidence of blood culture-confirmed symptomatic TF in all vaccine recipients of the intervention clusters, compared with control clusters.

SECONDARY OUTCOMES:
Safety Assessment | 3 years
  1) Proportion of adverse events in participants receiving Vi-TT compared with MCV-A, measured by:
  * The proportion of participants in each group of a sub-sample of the cohort developing adverse events/adverse reactions within the first 7 days post-vaccination.
  * The proportion of participants in each group of the cohort developing serious adverse events during the entire study period, as determined by self-reporting at follow-up contact.
Overall protection | 3 years
  The incidence of blood culture-confirmed symptomatic TF in all residents of the intervention clusters compared with that in all residents of control clusters
Total protection against severe typhoid. | 3 years
  The incidence of severe TF in vaccinated individuals in intervention clusters compared to control clusters
Total protection against clinical typhoid. | 3 years
  The incidence of clinical typhoid fever cases, defined as persistent fever (tympanic (≥38.0℃) or axillary temperature (≥37.5℃) or reported fever for ≥3 consecutive days) with abdominal complaints at a study surveillance site in vaccinated individuals in intervention clusters compared to control clusters.
Overall protection against clinical typhoid. | 3 years
  The incidence of clinical typhoid fever cases presenting at a study surveillance site among all residents of the Vi-TT clusters compared to the control vaccine clusters.
Indirect Protection aganist Blood Culture Confirmed Typhoid. | 3 years
  The incidence of blood culture-confirmed symptomatic TF in non-vaccinees of the intervention clusters compared with control clusters.
Seroconversion rates | 3 years
  The seroconversion rates as measured by enzyme linked immunosorbent assay (anti-Vi IgM and IgG) for S. Typhi and iNTS at defined time points in a age-stratified subset of intervention and control vaccinees.
Geometric mean titers | 3 years
  The antibody concentration as measured by enzyme linked immunosorbent assay (anti-Vi IgM and IgG) for S. Typhi and iNTS at defined time points in a age-stratified subset of intervention and control vaccinees.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Marks, PhD, Principal Investigator — University of Cambridge; Ellis Owusu Dabo, PhD, Principal Investigator — Kwame Nkrumah University of Science and Technology
Locations (1):
- Kwame Nkrumah University of Science and Technology, Kumasi, Ashanti Region, Ghana

IPD SHARING:
Plan to Share IPD: No
Sharing can be considered on a case-by-case basis considering the intended use and impact.